CLINICAL TRIAL: NCT01087632
Title: Effects of Armolipid Plus on Indices of Insulin Resistance in Patients With Metabolic Syndrome
Brief Title: Armolipid Plus and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rottapharm (Industry)
Collaborators: Federico II University (Other)
Responsible Party: Massimo D'Amato, MD, Rottapharm
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARMP-09
Record Dates: First submitted 2010-03-12; First posted 2010-03-16 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-09

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome Insulin-resistance Endothelial Function
MeSH Terms: conditions — Metabolic Syndrome | interventions — Berberine; red yeast rice; Lovastatin; policosanol; coenzyme Q10; astaxanthine; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Armolipid Plus (Experimental): Armolipid Plus is an association of berberine 500 mg, red yeast rice titled in 3 mg monacolin K,- policosanol 10 mg,coenzyme Q10 2 mg,astaxanthin 0,5 mg,folic acid 0,2 mg
  Interventions: Dietary Supplement: Armolipid Plus
- Placebo (Placebo Comparator): Placebo matching Armolipid plus
  Interventions: Dietary Supplement: Armolipid Plus

INTERVENTIONS:
Dietary Supplement: Armolipid Plus — Armolipid Plus 1 tablet QD for 18 weeks
  Other Names: berberine; red yeast rice; monacolin K; policosanol; coenzyme Q10; astaxanthin; folic acid

SUMMARY:
Metabolic syndrome is a highly prevalent condition characterized by visceral obesity, abnormalities of glucidic and lipid metabolism, and increased risk for cardiovascular events. Such findings appear to be associated with a decrease in insulin sensitivity. Management of metabolic syndrome is currently aimed at treating individual components of the disease without addressing this underlying pathophysiologic mechanism; this translates into multidrug regimens, high costs and patient compliance issues.

Armolipid Plus (an association of berberine 500 mg, red yeast rice titled in 3 mg monacolin K,policosanol 10 mg,coenzyme Q10 2 mg,astaxanthin 0,5 mg,folic acid 0,2 mg) has been found to be effective at reducing blood cholesterol and triglycerides, and at improving endothelial function; subgroup analyses also suggested a benefit on indices of insulin resistance.

Aim of the study is to evaluate the effects of Armolipid Plus on insulin sensitivity and on the diagnostic parameters of metabolic syndrome.

60 patients will be enrolled in this randomized, double-blind, placebo-controlled trial; active treatment will consist of Armolipid Plus (1 tbl qd).

Primary end point will be the reduction of the insulin/glucose ratio, both after overnight fast (HOMA index) and after an oral glucose tolerance test (OGTT).

ELIGIBILITY:
Inclusion Criteria:

Male and Female 18-65 aged, with diagnosis of metabolic syndrome, defined by the presence of waist circumference > 102 cm (M) or >88 cm(F), and two or more of these criteria:

* fasting blood glucose >100 mg;
* systolic blood pressure >135 or diastolic blood pressure >85 mmHg or patients in treatment with antihypertensive drugs;
* triglyceridemia >150 mg/dl;
* HDL cholesterolemia < 40 mg/dl(M), < 50 mg/dl(F).

Exclusion Criteria:

* pregnancy
* diabetes mellitus in pharmacologic treatment;
* hepatic failure;
* creatininemia >2 mg/dl;
* triglyceridemia > 500 mg/dl;
* heart failure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Insulin/glucose ratio after overnight fast | 18 weeks
  HOMA INDEX
Insuline/glucose ratio after an oralglucose tolerance test | 18 weeks
  OGTT

SECONDARY OUTCOMES:
BMI | 18 weeks
  evaluation of weight and BMI
Glycemia | 18 weeks
  Blood Glucose
Endothelial function | 18 weeks
  endothelial function assessed by Flow Mediated Dilation
C reactive protein. | 18 weeks
  dosage of CRP
Serum lipidemia | 18 weeks
  measure of TG and cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Serafino Fazio, MD, Principal Investigator — Federico II University
Locations (1):
- Federico II University - Department of Internal Medicine, Naples, Naples, Italy